CLINICAL TRIAL: NCT00487149
Title: Respiratory Muscle Strength in Bronchiectasis: Repeatability and Reliability
Status: Completed | Type: Observational
Sponsor: University of Ulster (Other)
Other Study IDs: 1233R0203
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Healthy; Bronchiectasis
Keywords: Repeatability; Respiratory Muscle Strength
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Respiratory muscle strength is used as an outcome measure in intervention studies. There are reference values for respiratory muscle strength in 'healthy' people but not in those with bronchiectasis disease. The aim of this study is to investigate the reliability of respiratory muscle strength measurements and identify reference values for those with stable moderate to severe bronchiectasis disease.

DETAILED DESCRIPTION:
Twenty 'healthy' participants and 20 participants with moderate to severe bronchiectasis in a stable state were recruited. Three readings for pulmonary function (FEV1); and respiratory muscle strength (PImax;PEmax) were taken on two occasions 10-14 days apart according to a standardised protocol.

A standard protocol and instructions for all measurements of respiratory strength were used. Measurements were made at the same time of day and with no change in medication. Before the subject undertook the respiratory muscle strength tests the assessor provided verbal explanations and demonstration of the procedure. The subject then had a practice run before values were recorded. Values were reported as positive numbers.

Measurements were obtained by one of three assessors. Pretraining ensured that all assessors followed standardised methodology.

Pulmonary function measures were conducted according to the ATS standards (ATS, 2002). The FEV1 percentage predicted value was reported as the ECCS scale. FEV1 had to remain within 10% to eliminate the possibility of a pulmonary exacerbation.

Respiratory muscle strength measurements were conducted using a handheld mouth pressure meter, a one way inspiratory or expiratory valve, a single use bacterial filter, nose clips and a standard flanged mouthpiece (Micro Medical Ltd UK). The pressure gauge was calibrated with a small air leak (greater than 1mm in diameter) to reduce use of the buccal muscles. A hand held mouth pressure machine computed average pressures in cmH2O sustained over two seconds and a microprocessor displayed a digital result.PImax was measured near residual volume after maximal expiration. PEmax was measured near total lung capacity after a maximal inspiration. There was a minute's rest between each manoeuvre. Verbal encouragement was given to each participant to obtain maximal effort. Three technically acceptable readings for inspiratory and expiratory pressure measured were recorded.

All participants gave written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* All participants:over 40 years of age,non smokers,able to perform lung function tests and available for a repeat measure 10-14 days later.
* Specific inclusion criteria for healthy participants:no known respiratory or cardiac condition and no prescription antibiotics for a chest complaint.
* Specific inclusion criteria for bronchiectasis group:

  * Diagnosis of bronchiectasis by CT scan;
  * Moderate to severe disease (FEV1 < 60% predicted);
  * In a stable state i.e. no administration of oral or intravenous antibiotics in preceding 3 weeks;
  * No change in medication such as bronchodilators, oxygen, long term prophylactic antibiotics or steroids in the 3 weeks preceding the study.

Exclusion Criteria:

* Any co-morbid condition that could influence muscle strength or if participants live greater than 50 miles from the hospital.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-10; Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fidelma Moran, BSc(Hons), Principal Investigator — University of Ulster
Locations (1):
- Belfast City Hospital, Belfast, Northern Ireland, United Kingdom

REFERENCES:
- [Derived] Moran F, Piper A, Elborn JS, Bradley JM. Respiratory muscle pressures in non-CF bronchiectasis: repeatability and reliability. Chron Respir Dis. 2010 Aug;7(3):165-71. doi: 10.1177/1479972310375595. PMID 20688894